CLINICAL TRIAL: NCT06255938
Title: Prevalence of HPV and HPV Vaccination Among Victims of Sexual Violence
Brief Title: Prevalence of HPV (Human Papilloma Virus) and HPV Vaccination Among Victims of Sexual Violence
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire Saint Pierre (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: B0762023230706
Record Dates: First submitted 2024-02-01; First posted 2024-02-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Human Papilloma Virus; Sexual Assault; Sex Abuse
MeSH Terms: interventions — Vaginal Smears

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Vaginal, anal and oral smears for testing HPV
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: smears — PCR smears for HPV testing will be performed

SUMMARY:
By a prospective single center cohort study in the Sexual Assault Care Center (SACC) of the CHU (Centre Hospitalier universitaire) Saint Pierre in Brussels, we would like to :

* to evaluate the prevalence of HPV infections in the population of women over 15 years old admitted for rape
* to determine the prevalence of HPV and the clearance in HPV-vaccinated and unvaccinated patients

DETAILED DESCRIPTION:
The investigators will conduct a prospective single center cohort study in the SACC of the CHU Saint Pierre in Brussels.

Population:

the investigators will include all women over 15 years admitted to the SACC of Brussels between 5/02/2024 and 05/02/2024 for rape (vaginal and/or oral and/or anal penetration) after signing the consent.

PCR (polymerase chain reaction) smears for HPV testing will be performed after obtaining consent from the victims. These smears will be performed at the oral, vaginal and anal site. The smears will be taken either by the patient or by the legal nurse, according to the victim's wishes. Ideally, 3 smears should be taken : oral, vaginal and anal.

It will be carried out at the same time as all other sexual transmitted deseases tests and should therefore not be perceived as more invasive or time-consuming.

These smears will be performed two times: at the first visit of the patients to the SACC and after 12 at 18 months.

Appointment reminders will be sent by phone contact.

The test used is a swab analyzed by PCR via the AML laboratory. They confirmed that this is the most sensitive method for detecting HPV in vaginal and anal areas, and probably also in oral areas.

The HPVs obtained via PCR are: 16 18 45 33 58 31 52 35 59 39 51 56 68 67 53 66 6 and 11. Results will therefore be classified as low-risk, high-risk or HPV-negative.

Patients will be notified if a high-risk HPV test is detected, and treatment will be offered depending on the type of follow-up required according to the international recommendations.

Outcomes:

* Define high-risk HPV carriage in the SACC population.
* Define the proportion of SACC patients vaccinated for HPV.

Secondary objectives:

* To characterize HPV subtypes, according to the type of assault and infected sites (vaginal-cervical, anal, oral).
* To determine the prevalence of HPV and the clearance in HPV-vaccinated and unvaccinated patients (itself assessed by the presence of one type of HPV in the first smear and its absence in the followed smears).

ELIGIBILITY:
Inclusion Criteria:

* women over 15 years admitted for rape speaking in french, dutch or english (and therefore able to sign an inform consent in french, dutch or english)

Exclusion Criteria:

* tourist or other people who will not in belgium one year after their first test

Min Age: 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Women admitted for sexual assault to the SACC (Sexual Assault Care Center) of the CHU Saint-Pierre of Brussel
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
to evaluate the prevalence of HPV infections in the population of women over 15 years victim of sexual assault | at the admission

SECONDARY OUTCOMES:
To characterize HPV subtypes, according to the type of assault and infected sites | at the admission
To determine the prevalence of HPV and the clearance in HPV-vaccinated and unvaccinated patients | at the admission and one year later

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Rousseau, Dr, Principal Investigator — Centre Hospitalier Universitaire Saint Pierre

IPD SHARING:
Plan to Share IPD: No